CLINICAL TRIAL: NCT00881374
Title: Study for Dermatological Evaluation of Topic Compatibility (Primary and Accumulated Dermic Irritability, Dermic Sensitivity) of Dermacyd Infantile (Lactic Acid).
Brief Title: Dermacyd Infantile (Lactic Acid)- Compatibility.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LACAC_L_04679
Record Dates: First submitted 2009-04-10; First posted 2009-04-15 (Estimated); Last update posted 2009-04-15 (Estimated); Status verified 2009-04

CONDITIONS: Hygiene

ARMS (1):
- Dermacyd Infantile (Lactic Acid) (Experimental): six weeks treatment
  Interventions: Drug: LACTIC ACID(ND)

INTERVENTIONS:
Drug: LACTIC ACID(ND) — Dermacyd Infantile (Lactic Acid)

SUMMARY:
Primary Objective:

To demonstrate the absence of irritation potential (primary dermic irritability and cumulated dermic irritability) and allergic potential (sensibilization) of the product Dermacyd Infantile.

ELIGIBILITY:
Inclusion criteria:

* Photo type Skin I,II, III e IV
* Integral skin test in the region
* Willingness in following the study procedures and to be present in the clinic at the days and scheduled time for medical evaluations and for application of occlusion.

Exclusion criteria:

* Lactation or gestation
* Use of Anti-inflammatory 30 days and/or immunosuppressant drugs during 3 months before the selection
* Diseases which can cause immunity decrease, such as HIV, diabetes
* Previous atopy
* History of sensitivity or irritation for topic products
* Active cutaneous diseases which can interfere in the study results
* Use of new drugs and/ or cosmetics during the study
* Cutaneous reactivity
* Previous participation in studies, which had used the product
* Volunteers who have immunodeficiency congenital or acquired
* Relevant clinical history or present evidence of alcohol abuse or others drugs
* Non tolerance to some component of the study product.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The absence of primary and accumulated dermic irritability and dermic sensitivity will be evaluated using International Contact Dermatitis Research Group (ICDRG) scale. | During 6 weeks (i.e. treatment period)

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil